CLINICAL TRIAL: NCT01584986
Title: Autologous Stem Cell Therapy for the Treatment of Patients With Peripheral Artery Disease
Brief Title: Autologous Angiogenic Cell Precursors (ACPs) for the Treatment of Peripheral Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Salus Ltd. (Industry)
Collaborators: TheraVitae Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACP_CLI_P01
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACP treated (Active Comparator): Autologous angiogenic cell precursors (ACPs) were injected into the ischemic gastrocnemius muscle in addition to the conventional treatment.
  Interventions: Biological: ACP injections
- Control (No Intervention): Control patients were treated with the conventional therapy.

INTERVENTIONS:
Biological: ACP injections — Peripheral blood-derived, ex vivo expanded autologous angiogenic cell precursors (ACPs)
  Arms: ACP treated

SUMMARY:
Regeneration of the occluded peripheral arteries by autologous stem cell therapy is an emerging treatment modality for no-option patients with peripheral artery disease (PAD). The purpose of this study was to assess safety and efficacy of ex vivo expanded, peripheral blood-derived, autologous angiogenic cell precursors (ACPs) in no-option PAD patients.

DETAILED DESCRIPTION:
Late-stage no-option PAD patients with a high risk of amputation of the affected limb were enrolled and randomized into treated and control groups. In the 10 ACP treated patients the stem cells were injected into the ischemic gastrocnemius muscle. The 10 control patients were treated with the conventional therapy. Physical examination, a treadmill walking test were performed, ankle brachial index (ABI), transcutaneous oxygen pressure (TcO2) were measured at baseline, 1 and 3 months later. Digital substraction angiography and SF-36 quality-of-life (QoL) questionnaire were also performed at baseline and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having one or more clinical indications diagnostic of CLI such as: distal extremity pain at rest that requires the subject to use analgesics for > 2 weeks; or peripheral ischemic ulcer(s); or areas of gangrene ; or non-healing ischemic ulcers; and
* Subjects having one or more of the following hemodynamic indicators of severe peripheral arterial occlusive disease: I. Ankle brachial index ≤ 0.45 or II. Toe brachial index ≤ 0.35 or III. TcPO2 / TcO2 of ≤ 40 mmHg.
* The subject being a poor candidate for standard revascularization treatment options for peripheral arterial disease, based on inadequate bypass conduit, or unfavorable anatomy;
* Age 18 to 80 years;
* Male or non-pregnant, non-lactating female;
* Informed consent obtained and consent form signed.

Exclusion Criteria:

* Patient having on angiography a meaningful supra-popliteal occlusion that may relate to symptoms of CLI;
* Subjects, who in the opinion of the investigator, have a vascular disease prognosis that indicates they would require a major amputation (at or above the ankle) within 4 weeks of start of treatment;
* Patient who received blood transfusions during the previous 4 weeks (to exclude the potential of non-autologous ACPs in the harvested blood);
* Inability to communicate (that may interfere with the clinical evaluation of the patient);
* Major operation during the preceding 3 months;
* Myocardial infarction or brain infarction or uncontrolled myocardial ischemia or persistent severe heart failure (EF< 25 %) during the preceding 3 months;
* Significant valvular disease or after valve replacement;
* After heart transplantation;
* Cardiomyopathy;
* Renal failure (creatinine > 2 mg/dl );
* Hepatic failure;
* Anemia (lower than 11 mg/dl hemoglobin for female and lower than 12 mg/dl for male);
* Abnormal coagulation tests [platelets, PT (INR), PTT];
* Stroke within the preceding 3 years;
* Malignancy within the preceding 3 years;
* Concurrent chronic or acute infectious disease;
* Severe concurrent medical disease (e.g., septicemia, HIV-1,2/HBV/HCV infections, poorly controlled insulin-dependent diabetes mellitus; HbAlc > 8% and proliferative retinopathy, systemic lupus erythematosus, multiple sclerosis, amyotrophic lateral sclerosis);
* Chronic immunomodulating or cytotoxic drugs treatment;
* Patients who have rectal temp. above 38.4 ºC for 2 consecutive days;
* Patient unlikely to be available for follow-up.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Safety | 3 months
  Evaluation the safety of ACPs intramuscular injection
Rest pain | 3 months
Pain-free walking distance | 3 months
Ulcer size | 3 months
Gangrene dimension and intensity | 3 months
Obtain evidence for improvement of tissue perfusion due to ACPs injection | 3 months

SECONDARY OUTCOMES:
Reduction of CLI patients hospitalization time | 3 months
Decrease CLI patient amputation rate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: György Acsády, DSc, Principal Investigator — Semmelweis University Department of Cardiovascular Surgery
Locations (2):
- Hungary (2):
  - Kelen Hospital, Budapest
  - Semmelweis University Department of Cardiovascular Surgery, Budapest